CLINICAL TRIAL: NCT03228368
Title: The Predicted Potential of Quantitative T Cell Repertoire(TCR) Analysis Using Next-generation Sequencing (NGS) in Anti-PD-L1 Treatment in Non Small Cell Lung（NSCLC) Cancer Patients
Brief Title: The Predicted Potential of Quantitative T Cell Repertoire(TCR) in Anti-PD-L1 Treatment in NSCLC Patients
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: First Affiliated Hospital of Zhejiang University (Other)
Collaborators: Hoffmann-La Roche (Industry); Geneplus-Beijing Co. Ltd. (Industry)
Responsible Party: Sponsor
Other Study IDs: TCR-1
Record Dates: First submitted 2017-06-28; First posted 2017-07-24 (Actual); Last update posted 2017-07-24 (Actual); Status verified 2017-03

CONDITIONS: Non-Small Cell Lung Cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — atezolizumab

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

GROUPS / COHORTS (1):
- Atezolizumab (MPDL3280): Atezolizumab 1200 milligrams (mg) will be administered via intravenous (IV) infusion on Day 1 of each 21-day cycle until disease progression, death, unacceptable toxicity, withdrawal of consent, or study termination by sponsor, whichever occurs first.
  Interventions: Drug: Atezolizumab (MPDL3280A)

INTERVENTIONS:
Drug: Atezolizumab (MPDL3280A) — anti-programmed death-ligand 1 (PD-L1) antibody

SUMMARY:
This study is designed to evaluate the predicted potential of quantitative T cell repertoire (TCR) of T cell receptor chains using next-generation sequencing (NGS) in the treatment of the anti-programmed death-ligand 1 (PD-L1) antibody atezolizumab in participants with locally advanced or metastatic NSCLC who have progressed during or following a platinum-containing regimen. Treatment may continue until disease progression or unacceptable toxicity.

ELIGIBILITY:
Inclusion Criteria:

* Histologically documented, locally advanced or metastatic NSCLC
* Representative formalin-fixed paraffin-embedded (FFPE) tumor specimens available or at least 12 unstained, freshly cut serial sections with associated pathology report that are evaluable for PD-L1 expression and epidermal growth factor receptor (EGFR) mutation status prior to enrollment, except for known sensitizing EGFR mutations in which case 10 unstained slides are required and there is no need for central testing of EGFR mutation status
* Disease progression during or following treatment with a prior platinum-containing regimen for locally advanced, unresectable, inoperable, or metastatic NSCLC, or disease recurrence within 6 months of treatment with a platinum-based adjuvant and/or neoadjuvant regimen or combined modality with curative intent
* Measurable disease per RECIST Version 1.1
* Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1
* Life expectancy greater than or equal to (>/=) 12 weeks
* Adequate hematologic and end organ function
* Agreement to remain abstinent or use contraceptive methods among women of childbearing potential or male partners of women of childbearing potential
* Recovery from all acute toxicities from previous therapy

Exclusion Criteria:

* Active or untreated central nervous system (CNS) metastases
* Spinal cord compression not definitively treated or not clinically stable
* Leptomeningeal disease
* Uncontrolled pleural or pericardial effusions or ascites requiring recurrent drainage
* Uncontrolled tumor-related pain
* Uncontrolled hypercalcemia
* Malignancies other than NSCLC within 5 years prior to randomization, except for those curatively treated with negligible risk of metastasis or death
* Pregnant or lactating women
* Significant cardiovascular, pulmonary, or autoimmune disease
* Severe infection or major surgery within 4 weeks, or antibiotic treatment within 2 weeks prior to randomization
* Prior treatment with or hypersensitivity to study drug(s) or related compounds
* Inability to discontinue strong cytochrome P450 (CYP) 3A4 inhibitors
* Prior allogeneic bone marrow or solid organ transplant
* Known PD-L1 expression status from other clinical studies
* Positive human immunodeficiency virus (HIV) or hepatitis B or C
* Receipt of a live attenuated vaccine within 4 weeks prior to randomization
* Treatment with systemic immunomodulators within 4 weeks or five half-lives (whichever is shorter) prior to randomization
* Treatment with systemic corticosteroids within 2 weeks prior to randomization

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients diagnosed of locally advanced or metastatic non small cell lung cancer progressed during or following treatment with a prior platinum-containing regimen and subsequently recevied atezolizumab.
Sampling Method: Non-Probability Sample
Enrollment: 10 (Estimated)
Dates: Start 2017-03-01 (Actual); Primary Completion 2018-03-01 (Estimated); Study Completion 2018-12-01 (Estimated)

PRIMARY OUTCOMES:
T cell repertoire | From Screening until disease progression, death, or loss to follow-up (up to approximately 3 years overall)
  Change of T cell receptor repertoire during Anti-PL-L1 treatment.

CONTACTS AND LOCATIONS:
Locations (1):
- The First Affiliated Hospital of College of Medicine, Zhejiang University, Hangzhou, Zhejiang, China